CLINICAL TRIAL: NCT03715725
Title: A Post-marketing Retrospective Non-interventional Study Using Nationwide Registries and Electronic Medical Records to Investigate the Real-life Effectiveness and Major Bleeding Complications of Oral Anticoagulants in Norwegian Non-valvular Atrial Fibrillation Patients
Brief Title: A Nationwide Observational Study Looking at Effectiveness and Bleeding Complications of NOACs vs. VKA in Non-valvular Atrial Fibrillation Patients.
Acronym: PROTECT-AF
Status: Terminated | Type: Observational
Why Stopped: After feasibility assessment and due to delays in data receipt study was terminated
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 19468
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Non-valvular Atrial Fibrillation
MeSH Terms: interventions — Rivaroxaban; apixaban; Dabigatran; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Registry cohort: Registries in Norway are nation-wide and provision of the information is mandatory, which eliminates the risk of both selection and re-call bias. The large and detailed dataset also makes it possible to adjust for other risk factors on which information is available.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939); Drug: Apixaban (Eliquis); Drug: Dabigatran etexilate (Pradaxa); Drug: Warfarin (Marevan)
- Electronic Medical Records (EMR) cohort: Patients with NVAF diagnosis will be identified through extraction of patient-level data from EMRs from a number of hospitals in Norway, in order to describe these patients more closely regarding their clinical characteristics that are not available in nation-wide registers (e.g., in-patient treatments, anthropometric data and laboratory test results).
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939); Drug: Apixaban (Eliquis); Drug: Dabigatran etexilate (Pradaxa); Drug: Warfarin (Marevan)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Administration according to clinical practice
Drug: Apixaban (Eliquis) — Administration according to clinical practice
Drug: Dabigatran etexilate (Pradaxa) — Administration according to clinical practice
Drug: Warfarin (Marevan) — Administration according to clinical practice

SUMMARY:
Using mandatory nationwide registries and possibly hospital electronic medical records in Norway, the researchers want to understand how well a group of drugs called "non-vitamin K antagonist oral anticoagulants" (rivaroxaban - Xarelto; apixaban - Eliquis; dabigatran - Pradaxa) works in patients with non-valvular atrial fibrillation (this is a condition when the heart beats irregularly) compared to another older drug, a vitamin K antagonist oral anticoagulants (warfarin) and how safe these drugs are. The primary objective of the study is to assess the occurence of an ischemic stroke (a condition when an artery that brings blood to the brain is blocked) and intracranial hemorrhage (a serious condition when a diseased blood vessel within the brain bursts).

ELIGIBILITY:
Inclusion Criteria:

Registry cohort (Cohort 1)

Cohort 1a:

* Age ≥18 at the date of first OAC (Oral Anti-Coagulants) dispensation (index date)
* Diagnosed with atrial fibrillation or flutter in the period 5-year pre-index period. Defined as ICD10 codes; I480 (paroxysmal AF), I481 (persisting AF), I482 (chronic AF), I483 (typical AF), I484 (atypical AF) or I489 (unspecified atrial fibrillation or flutter) as given by either NPR (Norwegian Patient Register) or as a OAC (warfarin, dabigatran, rivaroxaban or apixaban) dispensed on the reimbursement code for AF in NorPD (Norwegian Prescription Database) (ICD10 I48 or ICPC-2 K78)
* Dispensation of a first-time prescription for an OAC during the study period 1 January 2014 to 31 May 2018. This initiation of an OAC is the index event and requires that there is no previous prescription for any OAC in the preceding 365 days (counted from the date of the first dispensation backward to the end of OAC supply).

Cohort 1b:

* Age ≥18 at the beginning of the study period (1 January 2014).
* Diagnosed with atrial fibrillation or flutter prior or during the study period. Defined as ICD10 codes; I480 (paroxysmal AF), I481 (persisting AF), I482 (chronic AF), I483 (typical AF), I484 (atypical AF) or I489 (unspecified atrial fibrillation or flutter) as given by NPR.
* No dispensation of a prescription for an OAC (warfarin, dabigatran, rivaroxaban or apixaban) during the study period 1 January 2014 to 30 June 2018. The index event will be the beginning of the study period (1 January 2014) and requires that there is no previous prescription for an OAC in the preceding 365 days.

EMR cohort (Cohort 2):

* Age ≥18 at the date of first OAC dispensation (index date).
* Diagnosed with atrial fibrillation or flutter in the 5-year pre-index period defined as one of the following ICD10 codes in the EMRs obtained from the hospitals in the South-Eastern Health Region; I480 (paroxysmal AF), I481 (persisting AF), I482 (chronic AF), I483 (typical AF), I484 (atypical AF) or I489 (unspecified atrial fibrillation or flutter).
* Dispensation of a first-time prescription for an OAC (warfarin, dabigatran, rivaroxaban or apixaban) during the study period 1 January 2014 to 31 May 2018. This initiation of an OAC is the index event and requires that there is no previous prescription of any OAC in the preceding 365 days (counted from the date of the first dispensation backward to the end of OAC supply).

Exclusion Criteria:

* Valvular atrial fibrillation defined as presence of ICD10 codes in NPR; I05.2 mitral stenosis with insufficiency, I05.8 other mitral valve diseases (mitral (valve) failure), I342 (non-rheumatic mitral valve stenosis), Z952 (presence of prosthetic heart valve) and procedure codes FKD (prosthetic replacement of mitral valve), FKA (Repair of mitral valve for stenosis), FKB (Annuloplasty of mitral valve for insufficiency), FKC (Repair of mitral valve for insufficiency), FKW (Other operations on mitral valve) and FMD (replacement of aortic valve).
* Deep Venous Thrombosis (DVT) as defined by ICD10 codes I80 (Phlebitis and thrombophlebitis), Pulmonary Embolism (PE) as defined by ICD10 code I26 or I82 (other venous embolism and thrombosis), Other venous embolism and thrombosis within last 6 months before index date.
* Knee and/or hip replacement surgery (NCSP (Nordic Classification of Surgical Procedures) procedure codes; NGB, NGC, NFB or NFC) 5 weeks before index date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise all adult OAC naïve NVAF patients in Norway who filled a prescription for an OAC (rivaroxaban, apixaban, dabigatran, warfarin) in the study period, defined as from 1 January 2014 to 30 June 2018 (or later depending on availability of data) and followed until outcome of interest, the end of the study period or death. This initiation of an OAC is the index event and requires that there is no previous prescription dispensed for an OAC in the preceding 365 days (from end date of OAC supply to date of new OAC dispensation).
Sampling Method: Non-Probability Sample
Enrollment: 70000 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Ischemic stroke | Retrospective analysis from 1 January 2014 to 30 June 2018
  Ischemic stroke is defined by the following ICD10 (International Classification of Diseases) codes:
  I63x: Cerebral infarction
Intracranial hemorrhage | Retrospective analysis from 1 January 2014 to 30 June 2018
  Intracranial haemorrhage (ICH) is defined by the following ICD10 codes:
  I60x Subarachnoid haemorrhage I61x Intracerebral haemorrhage I62x Other non-traumatic intracranial haemorrhage

SECONDARY OUTCOMES:
Overall stroke | Retrospective analysis from 1 January 2014 to 30 June 2018
  Overall stroke is defined by the following ICD10 codes:
  I60x: Subarachnoid haemorrhage I61x: Intracerebral haemorrhage I62x: Other nontraumatic intracranial haemorrhage I63x: Cerebral infarction I64x: Stroke, not specified as haemorrhage or infarction
Systemic embolism | Retrospective analysis from 1 January 2014 to 30 June 2018
  Systemic embolism is defined by the following ICD10 codes:
  I74x: Arterial embolism and thrombosis
Myocardial infarction | Retrospective analysis from 1 January 2014 to 30 June 2018
  Myocardial infarction is defined by the following ICD10 codes:
  I21x: Acute myocardial infarction I22x: Subsequent myocardial infarction
All-cause mortality | Retrospective analysis from 1 January 2014 to 30 June 2018
Major bleeding | Retrospective analysis from 1 January 2014 to 30 June 2018
  As defined by Cunningham algorithm and Internation Society of Thrombosis and Hemostasis (ISTH) for EMR cohort.
Demographic characteristics | Retrospective analysis from 1 January 2014 to 30 June 2018
Clinical characteristics | Retrospective analysis from 1 January 2014 to 30 June 2018
  Age, gender, CHA2DS2-VASc and HAS-BLED score, bleeding history, concomitant medications and co-morbidities
Drug utilization patterns | Retrospective analysis from 1 January 2014 to 30 June 2018

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Norway